CLINICAL TRIAL: NCT01245205
Title: A Phase I Study of MK-2206 in Combination With Lapatinib in Refractory Solid Tumors Followed by Dose-Expansion in Advanced HER2+ Breast Cancer
Brief Title: Akt Inhibitor MK2206 in Combination With Lapatinib Ditosylate in Patients With Advanced or Metastatic Solid Tumors or Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02550; NCI-2011-02550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WCCC-CO-10904; CDR0000688912; CO10904 (Other: University of Wisconsin Hospital and Clinics); 8709 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — MK 2206; Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (Akt inhibitor MK2206 and lapatinib ditosylate) (Experimental): Patients receive Akt inhibitor MK2206 PO QOD for 28 days (35 days for course 1) and lapatinib ditosylate PO QD or BID on days 1-28 (days 9-35 for course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt inhibitor MK2206; Drug: lapatinib ditosylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of Akt inhibitor MK2206 and lapatinib ditosylate in treating patients with solid tumors or breast cancer that has spread to other places in the body. Akt inhibitor MK2206 and lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of MK-2206 (Akt inhibitor MK2206) in combination with lapatinib (lapatinib ditosylate) in adult subjects with advanced solid tumors. (Dose Escalation Cohort) II. To further evaluate the safety of MK-2206 in combination with lapatinib administered to patients with locally advanced and unresectable or metastatic human epidermal growth factor receptor 2 positive (HER2+) breast cancer, previously treated with trastuzumab. (Dose Expansion Cohort)

SECONDARY OBJECTIVES:

I. To determine the clinical activity of MK-2206 in combination with lapatinib administered to subjects with advanced solid tumors. (Dose Escalation Cohort) II. To describe the dose-limiting toxicities (DLTs) of combined MK-2206 and lapatinib. (Dose Escalation Cohort) III. To determine the safety of MK-2206 and lapatinib administered in combination. (Dose Escalation Cohort) IV. To determine the pharmacokinetic and pharmacogenomic profile of MK-2206 in combination with lapatinib. (Dose Escalation Cohort) V. To assess for target (HER2-phosphoinositide 3-kinase [PI3K]-protein kinase B [AKT] pathway) inhibition via peripheral blood mononuclear cells (PBMCs) in the dose escalation cohort. (Dose Escalation Cohort) VI. To determine the clinical activity of MK-2206 and lapatinib administered in combination to patients with locally advanced and unresectable or metastatic HER2+ breast cancer. (Dose Expansion Cohort) VII. To determine the progression-free rate following MK-2206 in combination with lapatinib when administered at the MTD level to subjects with HER2+ metastatic breast cancer (MBC). (Dose Expansion Cohort) VIII. To determine the pharmacokinetic and pharmacogenomic profiles of MK-2206 in combination with lapatinib. (Dose Expansion Cohort) IX. To assess for mechanisms of lapatinib resistance by evaluating tumor tissue for phosphatase and tensin homolog (PTEN) loss using immunohistochemistry. (Dose Expansion Cohort) X. To assess for mechanisms of lapatinib resistance by evaluating tumor tissue for oncogenic mutations in PI3K. Tumor response to combination therapy with lapatinib and MK-2206 will be correlated with presence/absence of PI3K activating mutations and PTEN loss. (Dose Expansion Cohort) XI. To assess for mechanisms of lapatinib resistance by assessing for target (HER2-PI3K-AKT pathway) inhibition via peripheral blood mononuclear cells (PBMCs). (Dose Expansion Cohort)

OUTLINE: This is a dose-escalation study.

Patients receive Akt inhibitor MK2206 orally (PO) every other day (QOD) for 28 days (35 days for course 1) and lapatinib ditosylate PO once daily (QD) or twice daily (BID) on days 1-28 (days 9-35 for course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and patients on the expanded cohort are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed advanced or metastatic solid tumor for which no standard curative measure exists
* Patients must have either evaluable or measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients may have previously had disease progression on lapatinib, but should not have demonstrated prior serious or life-threatening intolerance to doses of lapatinib exceeding 1000 mg per day
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (or Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< upper limit of normal (ULN); in the case of a patient with known Gilbert's disease, s/he will be eligible as long as total serum bilirubin is less than 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times upper limit of normal
* Creatinine =< ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 by Cockcroft-Gault for patients with creatinine levels above institutional normal
* Patients with treated, stable brain metastases are allowed to enroll; patients must be at least 4 weeks from radiation and off any medications used to treat brain metastases; patients are allowed to be on anti-epileptic medications that are not metabolized by cytochrome P450; patients with brain metastases must have stable brain imaging within 4 weeks prior to starting study

  * Patients with progressive brain metastases who are not candidates for further local therapy (e.g. more radiation or surgery) but who have clinically asymptomatic brain are also eligible to enroll, as long as predicted life expectancy with the brain metastases meets or exceeds study requirements
* Women of childbearing potential and men should use contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation AS WELL AS for one month after stopping use of the study agents

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* PART 2A: Patients must have histologically or cytologically documented locally advanced and unresectable OR metastatic breast cancer
* PART 2A: Patients must have HER2+ cancer as defined by either: (a) 3+ for HER2 by immunohistochemistry (IHC), or (b) fluorescence in situ hybridization (FISH) or in situ hybridization (ISH) mean locus-to-centromeric ratio greater than or equal to 2.2; these analyses must be determined on an invasive component of the cancer at either the primary site or the metastatic site
* PART 2A: Patients must have previously received trastuzumab, either in the adjuvant or metastatic setting
* PART 2A: All patients in this cohort must have archived primary or metastatic tissue blocks available

Exclusion Criteria:

* Patients who have had chemotherapy, therapy with trastuzumab, bevacizumab or other targeted therapy, or radiotherapy within 4 weeks (6 weeks for regimens including carmustine [BCNU], nitrosoureas or mitomycin C) prior to entering the study; the following will apply with regards to endocrine therapy:

  * Patients receiving an aromatase inhibitor (AI) are eligible as long as they stop the AI one day prior to beginning study agents
  * Patients receiving tamoxifen or fulvestrant should have received their last dose at least 2 weeks prior to beginning study agents
* Patients who have not recovered (=< grade 1) from adverse events due to agents administered more than 4 weeks earlier (tolerable grade 2 adverse events may be allowed at the discretion of the investigator)
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206, lapatinib or other agents used in the study
* Patients receiving any medications or substances that are strong or moderate inhibitors or inducers of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP 450 3A4) are ineligible unless they can be transitioned off this medication prior to study drug initiation

  * Patients on strong or moderate inhibitors/inducers will become eligible if they discontinue all such medications at least 5 days prior to start of therapy and no further doses are anticipated for the duration of investigational therapy

    * In order to be considered a contraindicated medication, a patient must be taking the drug systemically and on a regular and scheduled basis; for example, a topical medication taken intermittently need not be stopped
  * Patients currently taking weak CYP3A4 inducers, and/or inhibitors are eligible
  * Patients currently taking sensitive substrates with narrow therapeutic indices are ineligible unless:

    * The medication can be monitored clinically in the opinion of the principal investigator (PI)/Study Chair; monitoring will be performed on a schedule to be determined by the PI/study chair and treating physician (MD); for example, a substrate medication that can be clinically monitored is digoxin
    * If the medication CANNOT be monitored clinically, they discontinue all such medications at least 5 days prior to start of therapy and no further doses are anticipated for the duration of investigational therapy
* Patients with diabetes or at risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled before the patient enters the trial

  * Inadequately controlled diabetes mellitus or hyperglycemia will be defined as:

    * Hemoglobin A1c > 8%
    * Fasting blood glucose over 200
    * Diabetes which requires injected insulin
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* A baseline QT interval corrected by Fridericia's formula (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study; medications that may cause QTc interval prolongation should be avoided by patients entering on trial
* Patients with a left ventricular ejection function (LVEF) less than 50% or the lower limit of institutional normal are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with either MK-2206 or lapatinib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
MTD of Akt inhibitor MK-2206 and lapatinib ditosylate, defined as the dose level at which less than one-third of patients experience a DLT as graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.4 (Part I) | 35 days
Incidence of adverse reactions to Akt inhibitor MK2206 and lapatinib ditosylate in patients with advanced and unresectable or metastatic HER2+ breast cancer previously treated with trastuzumab as assessed by NCI CTCAE v. 4 (Part II) | Up to 4 years
  Possible adverse events will be reported in tabular format.

SECONDARY OUTCOMES:
Response rate (complete or partial response or stable disease) measured by Response Evaluation Criteria in Solid Tumors (RECIST) (Part I) | Up to 4 weeks
  Two-sided 95% confidence intervals for the proportions of subjects with a confirmed anti-tumor response will be computed.
Incidence of DLTs assessed by NCI CTCAE v. 4 (Part I) | Up to 4 weeks
  The toxicities observed will be summarized by type and severity using the most recent version of the NCI CTCAE v.4 terminology. Both the number and severity of toxicity and adverse events will be analyzed in descriptive manner and presented in tabular format.
Incidence of adverse events, graded using NCI CTCAE v. 4 (Part I) | Up to 4 weeks
  Possible adverse events will be reported in tabular format.
Response rates using RECIST guidelines (Part II) | Up to 4 years
  Responses will be summarized by means of descriptive statistics and frequency tables. Confidence intervals for the proportions of subjects with a confirmed anti-tumor response will be computed in the expansion cohort.
Disease progression using RECIST guidelines (Part II) | Up to 4 years
Progression-free survival (PFS) rates (Part II) | Up to 4 years
  PFS times will be presented in a tabular format. If enough events will be observed, a Kaplan-Meier curve will be displayed.
Pharmacokinetic (PK) parameters of Akt inhibitor MK-2206 in combination with lapatinib ditosylate (Part II) | Pre-dose, 0 and 30 minutes, 1, 2, 4, 6, 8, 12, and 24 hours on days 1, 9, and 15 of course 1, and day 1 of subsequent courses
  All PK parameters will be summarized by using means, standard deviations and ranges. PK parameters of patients with severe toxicities (grade >= 3) will be compared to PK parameters of patients with no severe toxicities using Wilcoxon's rank sum test. Given the exploratory nature of these analyses, no multiplicity adjustments will be made.
Quantitative expression of proteins in tumor specimens (Part II) | Baseline
  Expressions for total HER2, PTEN, and AKT will all be presented descriptively (mean, standard deviation, median, range) in tabular format and correlated with response or clinical benefit using regression models.
Oncogenic mutations in PI3K (Part II) | Baseline
  Genotypes will all be presented descriptively in tabular format and correlated with pharmacokinetics and clinical responses via regression models. PK data means and standard deviations will be summarized by genotype and compared using a series of pairwise two-sample t-tests. Genotype analyses are exploratory, hence no multiplicity adjustments will be made.
Change in PBMC counts (Part II) | Baseline to up day 1 of last course of treatment
  Paired t-tests will be used to compare baseline values to each PBMC assessment timepoint post-baseline. Means and standard deviations will be tabulated at each timepoint and for each dose level. Given the exploratory nature of these analyses, no multiplicity adjustments will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Amye Tevaarwerk, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin